CLINICAL TRIAL: NCT04903652
Title: A Prospective Phase Ⅱ Clinical Study of Pyrotinib Maleate Combined With Vinorelbine in the Treatment of HER2-positive Advanced Breast Cancer That Has Failed Trastuzumab Therapy
Brief Title: Pyrotinib Maleate Combined With Vinorelbine in the Treatment of HER2-positive Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-Pyrotinib-NVB
Record Dates: First submitted 2021-05-19; First posted 2021-05-26 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-01

CONDITIONS: HER2-positive Advanced Breast Cancer
MeSH Terms: interventions — Vinorelbine

STUDY DESIGN:
Intervention Model Description: Pyrotinib Maleate plus Vinorelbine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib plus Vinorelbine (Experimental)
  Interventions: Drug: Pyrotinib Maleate; Drug: Vinorelbine

INTERVENTIONS:
Drug: Pyrotinib Maleate — Pyrotinib p.o. 400 mg once daily
Drug: Vinorelbine — Vinorelbine p.o. 40 mg once every other day

SUMMARY:
This study is a single-center, single-arm, prospective phase II clinical study, which mainly evaluates the efficacy and safety of pyrotinib maleate combined with oral vinorelbine in the treatment of HER2-positive advanced breast cancer.

DETAILED DESCRIPTION:
The most important treatment for HER2-positive breast cancer is based on anti-HER2 targeted therapy, combined with chemotherapy or endocrine therapy. China's original new anti-HER2 targeted therapy drug, pyrotinib, has obtained rapid approval from the country for its outstanding phase II clinical trial efficacy. In patients enrolled in the phase II trial, pyrotinib has a significant effect, but the combination of pyrotinib and capecitabine significantly increases the adverse reactions of diarrhea. For this reason, there is a lack of research on other combination schemes of pyrotinib in HER2 advanced breast cancer. In the first-line treatment, the combination therapy (HN) of trastuzumab and vinorelbine has shown that it also has a synergistic effect with vinorelbine in anti-HER2 targeted therapy. It provides a good evidence-based basis for the trial design of pyrotinib combined with vinorelbine soft capsules. This phase II clinical study is specially designed for preliminary exploration.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients between 18 and 75 years old;
2. ECOG physical status score 0-2 points;
3. The expected overall survival period is not less than 12 weeks;
4. Pathologically confirmed HER2 expression-positive recurrent/metastatic breast cancer patients; the standard for HER2 expression positive is immunohistochemical staining (IHC) detection of HER2 3+ and/or fluorescent in situ hybridization (FISH) positive The researcher of the test center reviews and confirms).
5. The disease progresses during or after treatment with trastuzumab (stopping the drug for less than 12 months);
6. The number of chemotherapy lines used in the recurrence/metastasis stage is less than or equal to 2 lines;
7. Patients who have at least one measurable lesion [spiral CT scan ≥10 mm (CT scan thickness not greater than 5mm)] and who have progressed after or during the last anti-tumor treatment (RECIST version 1.1);
8. The main organs are functioning normally, that is, they meet the following standards:

1) The standard of routine blood examination should meet: Hb≥100 g/L (no blood transfusion within 14 days); ANC≥1.5×109 /L; PLT≥75×109 /L; 2) The biochemical inspection shall meet the following standards: TBIL≤1.5×ULN (upper limit of normal value); ALT and AST≤2.5×ULN; if there is liver metastasis, ALT and AST≤5×ULN; Serum creatinine ≤1.5×ULN, creatinine clearance ≥50ml/min (based on Cockroft and Gault formula); 3) Heart color Doppler ultrasound Left ventricular ejection fraction (LVEF) ≥50%; 9. For female patients who have not undergone menopause or have not undergone surgical sterilization: during treatment and at least 7 months after the last dose in the study treatment, agree to abstain from sex or use an effective method of contraception. 10. Patients voluntarily join this study, have good compliance with the planned treatment, understand the research process of this study, and sign written informed consent.

Exclusion Criteria:

1. There is fluid in the third space that cannot be controlled by drainage or other methods, such as pleural fluid and ascites;
2. There are many factors that affect the oral and absorption of drugs (such as inability to swallow, gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.);
3. Severe heart disease or discomfort, including but not limited to the following diseases:

   * Confirmed history of heart failure or systolic dysfunction (LVEF <50%)
   * High-risk uncontrolled arrhythmia, such as atrial tachycardia, resting heart rate> 100 bpm, significant ventricular arrhythmia (such as ventricular tachycardia) or higher grade atrioventricular block (ie Mobitz II second degree atrioventricular block or third degree atrioventricular block)
   * Angina pectoris that requires anti-angina pectoris medication
   * Clinically significant heart valve disease
   * ECG shows transmural myocardial infarction -Poor hypertension control (systolic blood pressure> 180 mmHg and/or diastolic blood pressure> 100 mmHg).
4. Those who have been confirmed to be allergic to the drug components of this program; have a history of immunodeficiency, including positive HIV testing, or have other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation.
5. Patients who are known to be pregnant or planning to become pregnant, or patients of gestational age who are unwilling to take effective contraceptive measures during the entire trial period;
6. Suffer from serious concomitant diseases, such as infectious diseases.
7. Other malignant tumors have occurred in the past 5 years, except for cured cervical carcinoma in situ and non-melanoma skin cancer;
8. Patients who have participated in other experimental studies within 30 days before the first dose of study drug is administered;
9. Patients judged by the investigator to be unsuitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Estimated 24 months
  From enrollment to progression or death (for any reason)

SECONDARY OUTCOMES:
Objective response rate (ORR) | Estimated 24 months
  Ratio of CR and PR in all subjects
Disease Control Rate (DCR) | Estimated 24 months
  Ratio of CR ,PR and SD in all subjects
Overall survival (OS) | Estimated 36 months
  From enrollment to death (for any reason)
Security (CTCAE 5.0) | From informed consent through 28 days following treatment completion
  Adverse events are described in terms of CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Chunfang Hao, PhD, Principal Investigator — Department of Breast Cancer Medical Oncology
Locations (1):
- Tianjin Cancer Hospital, Tianjin, China